CLINICAL TRIAL: NCT03695276
Title: Pulmonary Specialist-Health Coach Consult (PuSHCon) Model to Improve Access to Specialist Consultation and Receipt of Recommended Evidence-based Care for Vulnerable Patients With Chronic Obstructive Pulmonary Disease (COPD) and Asthma
Brief Title: Pulmonary Specialist-Health Coach Consult Model Study
Acronym: PuSHCon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R56HL143366-01 (NIH); R01HL143366 (NIH)
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: COPD Asthma
Keywords: Health coaching; COPD; Asthma; Access to specialty care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, with randomization at the individual level
Who Masked: Investigator
Masking Description: Investigators and the Data Safety Monitoring Board will receive data summaries that mask identification of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PuSHCon model (Experimental): A health coach will contact patients with poorly controlled asthma or COPD. The health coach will gather information from the patient and medical record and review the case with a pulmonary specialist. The specialist will provide recommendations to the primary care clinician based on the case review; the specialist may request an in-person patient visit if needed. The health coach will follow up with the primary care clinician and will support implementation of recommendations that the the primary care clinician accepts,
  Interventions: Behavioral: PushCon Model
- Usual care (Active Comparator): Patients with poorly controlled asthma or COPD will receive the standard of care, which usually means management within primary care. The study team will provide in-service sessions on COPD and asthma guidelines to primary care clinicians in both arms. As in standard practice, a primary care clinician may refer a patient for specialty consultation or diagnostic testing at any time.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PushCon Model — Pulmonary specialist consultation facilitated by a trained health coach, who will gather information from the patient and medical record prior to the consultation and will using health coaching skills to support implementation of recommended care.
  Other Names: Pulmonary specialist-health coach consultation model
  Arms: PuSHCon model
Behavioral: Usual care — The standard of care, which usually means management within primary care.
  Arms: Usual care

SUMMARY:
The Pulmonary Specialist-Health Coach Consultation (PuSHCon) study examines the implementation of health coach-assisted consultations to improve access to specialist care and implementation of specialist recommendations for patients with COPD, asthma, and asthma COPD overlap syndrome (ACOS) for low-income and vulnerable patients seen at public health clinics. Three hundred sixty (360) patients from ten clinics will be enrolled in the study and randomized at the individual level to receive health coaching or usual care; 180 patients will receive usual care and 180 patients will receive the PuSHCon model.

DETAILED DESCRIPTION:
While evidence-based care for chronic obstructive pulmonary disease (COPD) and asthma can substantially reduce disease burden and prevent emergency visits and hospitalizations, it is estimated that 55% of patients with COPD do not receive all recommended care and that less than 50% of patients with asthma are well controlled.

The proposed study will evaluate the effectiveness of a novel model for pulmonary specialist-health coach consultations (PuSHCon) in its ability to increase access to specialty recommendations and the provision of evidence-based care for patients with chronic obstructive pulmonary disease (COPD) and/or asthma receiving care at federally qualified health centers (FQHCs). The specific aims of the study are to compare the use of evidence-based care and of patient reported outcomes 4 months after the consultation. In addition, the study will evaluate the cost per patient in each model to determine the model's effectiveness in increasing access and lowering cost.

The first aim of comparing the use of evidence-based care will be measured as the proportion of guideline-based recommendations that are ultimately received by the patients. The secondary endpoint for this aim will be measured through the proportion of patients receiving guideline-concordant medications at 4 months after consultation compared to baseline.

The second aim of the study regarding patient-reported outcomes will be measured primarily through the change in COPD and/or asthma related quality of life measures from baseline to 4 months post consultation. The secondary measure for this aim will look at changes in COPD and/or asthma specific symptom scores.

The third aim of the study is to assess the impact of this model on access to care and cost of care. Access will be measured by tracking the number of patients who successfully complete a consultation per month. Costs will be determined by calculating time spent per patients, as well as by health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* At least 18 years of age
* Diagnosed with asthma or COPD
* Experiencing uncontrolled symptoms or exacerbations

Exclusion Criteria:

* Do not plan to attend primary care clinic for at least 3 months
* Already engaged in pulmonary specialty care (defined as at least one visit in last 12 months)
* Cognitive dysfunction that would prevent interaction with a health coach
* Not having a phone at which the participant can be reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Willard-Grace, MPH, Principal Investigator — University of California, San Francisco
Locations (11):
- United States (11):
  - St. Anthony Medical Clinic, San Francisco, California
  - Tom Waddell Urban Health Clinic, San Francisco, California
  - Potrero Hill Health Center, San Francisco, California
  - Family Health Center, San Francisco, California
  - Mission Neighborhood Health Center, San Francisco, California
  - Richard H. Fine People's Clinic (General Medicine Clinic), San Francisco, California
  - Maxine Hall Health Center, San Francisco, California
  - Ocean Park Health Center, San Francisco, California
  - Southeast Health Center, San Francisco, California
  - Castro Mission Health Center, San Francisco, California
  - Silver Avenue Family Health Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PuSHCon Model | Usual Care
Started | 165 | 163
Completed | 126 | 125
Not Completed | 39 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PuSHCon Model | Usual Care | Total
Number analyzed (Participants) | 165 | 163 | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years
  Years | 51.9 (13.6) | 53.1 (14.0) | 52.5 (13.8)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: "Other" category includes individuals identifying as a gender other than male or female, as well as individuals who preferred not to answer the question
  Participants
    Female | 118 | 128 | 246
    Male | 43 | 34 | 77
    Other | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 9 | 16
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 60 | 63 | 123
  White | 23 | 19 | 42
  More than one race | 12 | 6 | 18
  Unknown or Not Reported | 59 | 63 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 56 | 115
  Not Hispanic or Latino | 106 | 107 | 213
  Unknown or Not Reported | 0 | 0 | 0
Breathing-related quality of life [Mean (Standard Deviation); unit: Scores on a scale] — St. George Respiratory Questionnaire Score (0-100, where 0 is best)
  Scores on a scale | 51.6 (16.6) | 52.0 (16.8) | 51.8 (16.7)

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Recommended Care
Description: Numerator: Number of guideline-based recommendations implemented by the patient; Denominator: Number of minimal recommendations based on GOLD/GINA guidelines
Time Frame: 16 weeks after enrollment
Measure: Mean (95% Confidence Interval); unit: Percentage of guidelines implemented
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 165 | 163
Percentage of guidelines implemented | 38.2 [31.3 to 46.6] | 23.7 [18.7 to 30.0]

2. Primary Outcome: Receipt of Recommended Medications
Description: Numerator: Number of people receiving all minimal recommended medications based on GOLD/GINA guidelines; Denominator: Number of people enrolled in study
Time Frame: 16 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 165 | 163
Participants | 126 | 110

3. Secondary Outcome: Provider Acceptance of Recommended Care
Description: Number of guideline-based recommendations where provider took action (e.g., prescribed or referred patient for care); Denominator: Number of minimal recommendations based on GOLD/GINA guidelines
Time Frame: 16 weeks after enrollment
Population: Number of recommendations accepted out of those provided
Measure: Count of Units; unit: Recommendations
Units Other Than Participants: Recommendations
Groups:
- Recommendations Made: Number of recommendations made by pulmonary specialist
Arm/Group | Recommendations Made
Number analyzed (Participants) | 165
Number analyzed (Recommendations) | 2824
Recommendations | 2425

4. Secondary Outcome: Patient-Reported Disease-specific Quality of Life (for Asthma and COPD) - Overall Score
Description: Score on St. George's Respiratory questionnaire (overall) with range of 0-100, where 0 is highest quality of life and 100 is lowest. (Full scoring manual located at: http://www.healthstatus.sgul.ac.uk/SGRQ_download/sgrq-c-manual-april-2012.pdf)
Time Frame: 16 weeks after enrollment
Population: Includes individuals who completed the 16 week survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 124 | 125
Scores on a scale | 37.6 (18.6) | 50.8 (18.2)

5. Secondary Outcome: Medication Adherence
Description: Number and percentage of patients taking all controller inhalers as prescribed for at least 5 of the last 7 days
Time Frame: 16 weeks after enrollment
Population: Includes individuals who completed the 16 week survey and reported taking a controller medication at the time
Measure: Count of Participants; unit: Participants
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 98 | 89
Participants | 48 | 42

6. Secondary Outcome: Patient-reported Quality of Care
Description: Mean score on Patient Assessment of Chronic Illness Care (PACIC) measure, with response options ranging from 1 (Almost never) to 5 (Almost Always). The scale is scored as an overall mean (1-5), with higher scores indicating a more frequent presence of high quality care. Four PACIC subscales (patient activation, delivery system practice design, goal setting/tailoring, problem solving/contextual), plus follow up/coordination are also represented by means of respective items.
Time Frame: 16 weeks after enrollment
Population: Includes individuals who completed the 16 week survey
Measure: Mean (Standard Deviation); unit: 1-5 Likert Scale (5 best)
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 118 | 122
1-5 Likert Scale (5 best) | 3.37 (1.11) | 3.12 (1.12)

7. Secondary Outcome: Disease Specific Symptoms Score (COPD & Asthma)
Description: Score on St. George's Respiratory questionnaire (symptom subscale) with range of 0-100, where 0 is highest quality of life and 100 is lowest. (Full scoring manual located at: http://www.healthstatus.sgul.ac.uk/SGRQ_download/sgrq-c-manual-april-2012.pdf)
Time Frame: 16 weeks after enrollment
Population: Includes individuals who completed a 16 week survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 114 | 122
Scores on a scale | 40.8 (21.1) | 49.7 (21.2)

8. Secondary Outcome: Proportion of Patients Who Engaged in Chronic Lung Disease Education
Description: Numerator: Number of people who engage with at least one existing resources such as group education classes or pulmonary care; Denominator: Number of people enrolled in the study
Time Frame: 16 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | PuSHCon Model | Usual Care
Number analyzed (Participants) | 165 | 163
Participants | 126 | 91

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | PuSHCon Model | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/163
Other Adverse Events (participants affected / at risk) | 0/165 | 0/163

LIMITATIONS AND CAVEATS:
The PuSHCon study randomized participants at the individual rather than the clinician or practice level.

This study was carried out in safety net practices within a single city and over a short duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT03695276/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03695276/ICF_001.pdf